CLINICAL TRIAL: NCT06067217
Title: Comparative Study of Tranexamic Acid, Estrogen for Treatment Abnormal Uterine Bleeding in Depot-medroxyprogesterone Acetate Users. A Randomized Controlled Trial
Brief Title: Comparative Study of Tranexamic Acid, Estrogen for Treatment AUB in DMPA Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 166/2566
Record Dates: First submitted 2023-09-13; First posted 2023-10-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-08

CONDITIONS: Abnormal Uterine Bleeding; Tranexamic Acid; Estrogen; Depot Medroxyprogesterone Acetate
Keywords: AUB; DMPA; Tranexamic acid; Estrogen
MeSH Terms: conditions — Metrorrhagia | interventions — Tranexamic Acid; Tablets; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Drug in concealed envelop which participant and care provider aren't see
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic acid (Experimental): Tranexamic acid 250 mg oral three times/day
  Interventions: Drug: Tranexamic acid 250 mg oral tablet
- Progynova (Experimental): Progynova 1 mg oral three times/day
  Interventions: Drug: Progynova 1 mg oral tablet

INTERVENTIONS:
Drug: Tranexamic acid 250 mg oral tablet — Compare between tranexamic acid and progynova to stop abnormal uterine bleeding in DMPA users
  Arms: Tranexamic acid
Drug: Progynova 1 mg oral tablet — Compare between tranexamic acid and progynova to stop abnormal uterine bleeding in DMPA users
  Arms: Progynova

SUMMARY:
Abnormal uterine bleeding is the most common problems to discontinue Depo-medroxyprogesterone acetate (DMPA) in Thailand. This clinical trial use to provide drug to stop abnormal uterine bleeding from DMPA

DETAILED DESCRIPTION:
Abnormal uterine bleeding is the most common problems to discontinue Depo-medroxyprogesterone acetate (DMPA) in Thailand. After discontinue DMPA, patients have not used any method. Unwanted pregnancy are rising. The reason of abnormal uterine bleeding from DMPA aren't clearly understand. In present, no standard treatment to treat abnormal utrerine bleeding in DMPA users.This clinical trial use to provide drug to stop abnormal uterine bleeding from DMPA with minimal dose and minimal side effect

ELIGIBILITY:
Inclusion Criteria:

* Abnormal uterine bleeding more than 7 days after first DMPA injection
* Provide inform consent with patient
* Can understand thai language

Exclusion Criteria:

* Have contraindication to use Tranexamic acid and estrogen such as hypertension, Stroke, MI, DM, Renal disease, Liver disease, CA breast etc.
* Have pathology in uterus from pelvic examination, pap smear and ultrasound
* Current pelvic infection
* Postpartum less than 6 months
* History deep vein thrombosis
* Breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Day to stop abnormal uterine bleeding between groups after receiving Tranexamic acid and estrogen | 1 week after intervention
  To Compare day to stop abnormal uterine bleeding between groups after receiving Tranexamic acid and estrogen

SECONDARY OUTCOMES:
Side effect after receiving Tranexamic acid | 1 week after intervention
  To study side effect after receiving Tranexamic acid
Side effect after receiving estrogen | 1 week after intervention
  To study side effect after receiving estrogen
Frequency of bleeding after DMPA injection | after DMPA injection
  To study frequency of bleeding after DMPA injection

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Krittiporn Mahachiraphat, Bangkok, Ratchathewi
  - Krittiporn Mahachiraphat, M.D., Phaya Thai, Ratchathewi

IPD SHARING:
Plan to Share IPD: No